CLINICAL TRIAL: NCT01604590
Title: Imaging Biomarkers of Tissue Microstructure and Vasculature as Predictors of Glioblastoma Multiforme Response to Treatment With Bevacizumab for Progressive Disease
Brief Title: Imaging Biomarkers of Tissue Microstructure and Vasculature as Predictors of Glioblastoma Multiforme
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 101652, MUSC
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-03

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Imaging Biomarkers; Bevacizumab; MRI
MeSH Terms: conditions — Glioblastoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- glioblastoma patients on bevacizumab
  Interventions: Radiation: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Radiation: Magnetic Resonance Imaging (MRI) — Magnetic Resonance Imaging (MRI) will be used to compare bevacizumab to the images of vessel and tumor structure.

SUMMARY:
This study is for subjects with a diagnosis of a brain tumor called glioblastoma that is being treated with bevacizumab. This study will use a new MRI technique to compare the images of blood vessels and tumor structure to the effectiveness of bevacizumab.

DETAILED DESCRIPTION:
This study is for subjects with a diagnosis of a brain tumor called glioblastoma that is being treated with bevacizumab. Bevacizumab is a drug that your doctor believes is the best treatment option available to subjects at this time for this type of tumor. Bevacizumab affects the growth of blood vessels by tumors such as glioblastoma, thus effectively starving the tumor of oxygen and food.

Magnetic Resonance Imaging (MRI) is a test done by a machine in the radiology department that takes pictures of your body using special magnets, rather than X-rays. With a new MRI scan technique the investigators can take very, very detailed images of the vessel and tumor structure. This project will allow us to compare the images of vessel and tumor structure to the effectiveness of Bevacizumab as a treatment option. With this project the investigators will hopefully develop an accurate way to predict whether or not Bevacizumab will be an effective treatment option for patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years of age
* Progressive glioblastoma patients who have been planned to receive bevacizumab
* Karnofsky Performance Status 50 or above (vd. Appendix A)
* Established pathologic diagnosis of glioblastoma
* Prior treatment with radiation and chemotherapy
* Neuroimaging progression of glioblastoma
* Able and willing to provide informed consent (or consent of a guardian)

Exclusion Criteria:

* Contraindication to MRI
* Contraindication to bevacizumab therapy
* Concurrent enrollment in other neuroimaging trials
* Prior therapy with bevacizumab
* Known hypersensitivity to MRI contrast
* Females who are nursing or pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects, 18-80 years old with progressive glioblastoma who receive bevacizumab
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
MRI to show differences between bevacizumab responses | 1 month
  The MRI parameters will help show the differences between bevacizumab-responsive and bevacizumab non-responsive recurrent glioblastoma

SECONDARY OUTCOMES:
Progression Free Survival at 3 months | 3 months
  The progression of the subject's disease will be evaluated at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Giglio, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States